CLINICAL TRIAL: NCT06861751
Title: Correlation Between Smart Phone Overuse, Craniovertebral Angle, Cervical Muscle Endurance and Temporomandibular Proprioception in Adolescents
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Zidan Ahmed Zidan, principal investigator, Cairo University
Other Study IDs: Mohamed-005616
Record Dates: First submitted 2025-03-01; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Smart Phone Addiction; Craniovertebral Angle; Temporomandibular Proprioception; Adolescents

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The study was done to:

1. Investigate the correlation between smart phone overuse and craniovertebral angle in adolescents.
2. Investigate the correlation between smart phone overuse and cervical muscle endurance in adolescents.
3. Investigate the correlation between smart phone overuse and temporomandibular joint proprioception in adolescents.

DETAILED DESCRIPTION:
This study was aimed to clarify the correlation between prolonged use of spinal traction on cervical curvature, muscle endurance, and temporomandibular joint proprioception in adolescents. It assisted physiotherapists in detecting and treating problems caused by prolonged spinal traction use, providing necessary precautions and treatments to prevent or alleviate this issue.

ELIGIBILITY:
Inclusion Criteria:

1. Both genders will be included.
2. Adolescents with age ranging from 17 to 19 years.
3. Adolescents using smart phone daily for not less than 4 years for 4 years.
4. All participants will be free from any medical disease, visual or hearing problem.
5. No history of temporomandibular joint complaints or disorder.

Exclusion Criteria:

1. Adolescent who cannot understand or follow instructions.
2. Congenital or acquired spinal deformities.
3. Adolescents with obesity.
4. Athlete adolescents.
5. Any neck or upper extremity Injury.
6. Neurological, musculoskeletal, and cardiopulmonary disease.
7. Adolescent with teeth braces during last 4 years

Ages: 17 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 160 adolescent from both sexes with their age ranging from 17 to 19 years and were smart phone addictors for not less than 4 years old
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of body mass index | at baseline
  A weight-height scale was used to measure the weight and height of each participant in both groups to calculate body mass index.

SECONDARY OUTCOMES:
Assessing the craniovertebral angle using software program | at baseline
  The study involves capturing a lateral view photo of a child's craniovertebral angle using reflective dots on the tragus and spinous process of the 7th cervical vertebrae. The camera is placed 1.5 meters away from the subject's shoulder level without rotation or tilt. The photographs are then transferred to a computer using software to assess the craniovertebral angle, which is defined as forward head posture with a craniovertebral angle of less than 50º.
Testing of temporomandibular joint Proprioception | at baseline
  Participants were given detailed instructions on assessment procedures, with a therapist standing in front of them at the same head level. Temporomandibular joint proprioception was measured using the Vernier caliper in all directions, including mouth opening, protrusion, and lateral jaw movements.
Measuring the Endurance of deep neck flexor muscles | at baseline
  The study involves a 20-pressure biofeedback device inflated to a baseline of 20 mmHg, followed by verbal feedback from the examiner. The subject performs neck flexion movements at different pressure levels (22, 24, 26, 28 and 30 mmHg) with 10 seconds hold at each level and 30 seconds rest between each level. The testing is terminated if the subject cannot hold 10 seconds at specific pressure levels or reaches a maximum level of 30 mmHg.

CONTACTS AND LOCATIONS:
Locations (1):
- out-patient clinic, faculty of physical therapy, Delta University for Science and Technology, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No